CLINICAL TRIAL: NCT03295773
Title: Morphologic Evolution and Remodeling of Intracranial Atherosclerosis: A Longitudinal Study by 3D-rotational Angiography
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Leung Wai Hong Thomas, Professor, Chinese University of Hong Kong
Other Study IDs: crec no. 2015.623
Record Dates: First submitted 2017-09-20; First posted 2017-09-28 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Ischemic Stroke; Atheroscleroses, Cerebral
Keywords: Ischemic Stroke; 3D-rotational angiography; Morphology; Atherosclerosis
MeSH Terms: conditions — Ischemic Stroke; Intracranial Arteriosclerosis; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Symptomatic stroke patient: Patients who are found signal void in a relevant intracranial internal carotid artery or middle cerebral artery (stenosis >60%) will proceed to a 3-Dimensional rotational angiography (3DRA) at baseline and in 12 months. All recruited patients will receive dual antiplatelet agents for 4 weeks, followed by aspirin alone. The investigator or neurologists shall regularly review the patients and treat the conventional cardiovascular risk factors based on four pre-specified goals, for example, LDL <1.8, HbA1c <6.0, blood pressure <140/90 and no smoking. The morphologic changes of the cerebral plaques with the intensity of the risk factor control in pre and post will be correlated.
  Interventions: Diagnostic Test: 3DRA

INTERVENTIONS:
Diagnostic Test: 3DRA

SUMMARY:
This study is to elucidate the morphologic evolution and remodeling of ICAD under stringent control of cardiovascular risk factors.

DETAILED DESCRIPTION:
The investigator has conducted extensive research on ICAD by transcranial Doppler ultrasound, CT angiography and perfusion studies, magnetic resonance imaging (MRI) and digital subtraction angiography (DSA) respectively. Currently, the investigator applied 3-dimensional rotational angiogram (3DRA), a selective intra-arterial catheter-based imaging technique that had a superior spatial resolution compared with CT, MRI or DSA in depicting minute (<3mm) angio-architecture. Through 3DRA, the investigator could appreciate the ICAD patho-anatomy from a near-infinite number of planes, analyzing the stroke mechanisms and morphological changes with much improved precision. A neuro-radiologist and a stroke neurologist blind to time sequence will measure the geometric parameters and the luminal narrowing by WASID method.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 30 to 85 years of age, inclusive.
2. Patients who have an acute infarct in diffusion-weighted MRI compatible with artery-to-artery thrombo-embolism and a relevant intracranial atherosclerotic stenosis ≥60%.
3. Patient who has no contra-indication for the proposed imaging tests.
4. Patient understands the purpose and requirements of the study, and has provided an informed consent.

Exclusion Criteria:

Patient with any of the following conditions would be excluded:

1. Stroke etiology uncertain or unrelated to intracranial atherosclerosis, such as cardioembolism, Moyamoya disease, small vessel disease or primary angiitis of CNS.
2. A tandem stenosis >50% at extra-cranial internal carotid artery.
3. Bleeding propensity: active peptic ulcer disease, major systemic hemorrhage within 30 days, thrombocytopenia (platelets <100 x 109/L), coagulopathy (INR >1.5).
4. A medical condition that would not allow the patient to adhere to the protocol or complete the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have acute cerebral ischemic symptoms attributed to a high-grade (≥60%) stenosis at a middle cerebral artery or intracranial segment of an internal carotid artery (ICA) would be reviewed by neurologists. If their stroke etiology and relevance to ICAD based on clinical syndrome, vascular imaging features and concurrent cardiovascular risks are eligible, they would be invited to join the study.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2016-08-22 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Morphologic Evolution and Remodeling of Intracranial Atherosclerosis | Dec, 2019
  The 3DRA images (the disparity in morphological attributes, including surface outline, angulations, plaque volume and distribution) of the patients in pre and post 12 month follow-up would be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wai Hong LEUNG, FRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No